CLINICAL TRIAL: NCT04399135
Title: Accuracy of Pulp Sensibility Test on Teeth With Deep Periodontal Pocket
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Bader Alharbi, Principal Investigator, Qassim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: # EA/F-2019-3005
Record Dates: First submitted 2020-05-09; First posted 2020-05-22 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis, Localized Aggressive; Periodontal Diseases; Endodontic Disease; Endodontic Inflammation; Periodontal Pocket; Periodontal Inflammation; Periodontal Attachment Loss; Periodontal Bone Loss; Periodontitis
Keywords: Periodontitis; Endodontic; Endo ice; Electric Pulp Tester (EPT).
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Dental Pulp Diseases; Pulpitis; Periodontal Pocket; Periodontal Attachment Loss; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: All patients who need root canal treatment would be screened to determine the periodontal condition for possible involvement in this study. They would be grouped into two groups, normal and periodontitis Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Patients (Active Comparator): All patients admitted to Qassim dental clinics, who need root canal treatment would be screened for possible involvement in this study
  Interventions: Diagnostic Test: Orthopantomogram X-ray view; Diagnostic Test: Endo-Ice; Diagnostic Test: Electric Pulp Tester (EPT)
- Periodontitis Patients (Active Comparator): All patients who need root canal treatment would be screened to determine the periodontal condition for possible involvement in this study. the periodontitis patients would be categorized according to the new periodontitis classification 2017 world workshop.
  Interventions: Diagnostic Test: Orthopantomogram X-ray view; Diagnostic Test: Endo-Ice; Diagnostic Test: Electric Pulp Tester (EPT)

INTERVENTIONS:
Diagnostic Test: Orthopantomogram X-ray view — taking an X-ray to determine bone loss level and attachment loss level for periodontitis classification
Diagnostic Test: Endo-Ice — Included teeth will be dried with 4x4 gauze then tested with a cold test using Endo-Ice.
Diagnostic Test: Electric Pulp Tester (EPT) — Included teeth will be dried with 4x4 gauze then tested with an Electric test using electric pulp tester (EPT).

SUMMARY:
The aim of this study is to evaluate the accuracy of pulp test in teeth presenting with deep periodontal pocket. The null hypothesis is no significant effect of periodontitis on the accuracy of pulp test.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the accuracy of pulp test in teeth presenting with deep periodontal pocket.

All patients who need root canal treatment would be screened to determine the periodontal condition for possible involvement in this study. They would be grouped into two groups, normal and periodontitis Group.

Included teeth will be dried with 4x4 gauze then tested with a cold test using Endo-Ice and electric pulp tester (EPT). Similar or adjacent teeth with no caries, restorations, or a history of the previous injury will be used as controls for that patient.

Upon accessing the tooth, no bleeding was counted as necrotic and any presence of blood was counted as a vital pulp

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 40 years old.
* Periodontitis grade II, III and IV
* Non-traumatized teeth.
* No prior non-surgical root canal treatment (NS RCT).

Exclusion Criteria:

* Periodontitis grade I.
* Patients with medically compromising conditions (ASA III and above).
* Trauma within the last six months.
* Partially necrotic pulps.
* Previously endodontically treated or initiation of treatment will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-02-25 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Is deep periodontal pocket affects pulp response, therefore, affects the accuracy of pulp test using "thermal" test? | through study completion, an average of 10 months.
  Endo-Ice would be used as a thermal test and participants will be asked to lift their hand up if they felt cold and keep it raised until the sensation is gone. Upon accessing the tooth, no bleeding would be counted as necrotic and any presence of blood counted as a vital pulp.
Is deep periodontal pocket affects pulp response, therefore, affects the accuracy of pulp test using "electrical" test? | through study completion, an average of 10 months.
  For Electrical Pulp tester (EPT) would be used as electrical pulp test. Any response before 80 was recorded as positive. Upon accessing the tooth, no bleeding would be counted as necrotic and any presence of blood counted as a vital pulp.

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University, Medical City, Dental Clinics, Buraidah, Al-Qassim Region, Saudi Arabia

REFERENCES:
- [Background] Bender IB. Reversible and irreversible painful pulpitides: diagnosis and treatment. Aust Endod J. 2000 Apr;26(1):10-4. doi: 10.1111/j.1747-4477.2000.tb00144.x. PMID 11359291
- [Background] Rotstein I, Simon JH. Diagnosis, prognosis and decision-making in the treatment of combined periodontal-endodontic lesions. Periodontol 2000. 2004;34:165-203. doi: 10.1046/j.0906-6713.2003.003431.x. No abstract available. PMID 14717862
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Result] Villa-Chavez CE, Patino-Marin N, Loyola-Rodriguez JP, Zavala-Alonso NV, Martinez-Castanon GA, Medina-Solis CE. Predictive values of thermal and electrical dental pulp tests: a clinical study. J Endod. 2013 Aug;39(8):965-9. doi: 10.1016/j.joen.2013.04.019. Epub 2013 May 21. PMID 23880259
- [Result] Jespersen JJ, Hellstein J, Williamson A, Johnson WT, Qian F. Evaluation of dental pulp sensibility tests in a clinical setting. J Endod. 2014 Mar;40(3):351-4. doi: 10.1016/j.joen.2013.11.009. Epub 2013 Dec 15. PMID 24565651
- [Result] Velitchka Dosseva, Antoaneta Mlachkova and Angela Gusiyska. Evaluation of The Pulp Vitality in Patients With Periodontitis/ Journal of IMAB - Annual Proceeding (Scientific Papers) 2007, vol. 13, book 2, pp.19-20

DOCUMENTS (1):
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT04399135/ICF_000.pdf